CLINICAL TRIAL: NCT00510432
Title: Inzidenz Und Art Heparin-induzierter Hautveränderungen
Brief Title: Incidence and Nature of Heparin-induced Skin Lesions in Medical Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Dr. Marc Schindewolf, Johann Wolfgang Goethe University Hospitals
Other Study IDs: 16/07
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Allergy
Keywords: heparin; heparin-induced thrombocytopenia; HIT; allergy; skin; dermatology; DTH; delayed-type hypersensitivity; histology; Patients receiving sc heparin therapy; Age over 18 years; Recruitment will stop when 20 patients with skin lesions are included
MeSH Terms: conditions — Hypersensitivity; Hypersensitivity, Delayed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- s.c. anticoagulant therapy: All patients with s.c. anticoagulant therapy (UFH, LMWH, heparinoids, fondaparinux)

SUMMARY:
An increased number of patients with heparin-induced skin lesions is reported in the literature. Heparin-induced skin lesions may result from either occlusion of cutaneous vessels in patients suffering from autoimmune HIT or from a type IV allergic reaction (delayed type hypersensitivity (DTH) response). However, the incidence and nature of heparin-induced skin lesions has not been determined in a prospective investigation.

To address this open issue is the goal of this ongoing, so far monocenter, clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 Y.
* s.c. anticoagulant therapy >6 days

Exclusion Criteria:

* history of HIT
* history of DTH to heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving s.c. anti-coagulation
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2007-04; Study Completion 2009-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ralf J Ludwig, MD, Principal Investigator — Department of Dermatology - Clinic of the Johann Wolfgang Goethe University
Locations (1):
- Department of Dermatology - Clinic of the Johann Wolfgang Goethe University, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Jappe U. Allergy to heparins and anticoagulants with a similar pharmacological profile: an update. Blood Coagul Fibrinolysis. 2006 Nov;17(8):605-13. doi: 10.1097/01.mbc.0000198992.18384.5a. PMID 17102645
- [Background] Ludwig RJ, Schindewolf M, Utikal J, Lindhoff-Last E, Boehncke WH. Management of cutaneous type IV hypersensitivity reactions induced by heparin. Thromb Haemost. 2006 Nov;96(5):611-7. PMID 17080218
- [Background] Bircher AJ, Harr T, Hohenstein L, Tsakiris DA. Hypersensitivity reactions to anticoagulant drugs: diagnosis and management options. Allergy. 2006 Dec;61(12):1432-40. doi: 10.1111/j.1398-9995.2006.01227.x. PMID 17073874
- [Background] Ludwig RJ, Schindewolf M, Alban S, Kaufmann R, Lindhoff-Last E, Boehncke WH. Molecular weight determines the frequency of delayed type hypersensitivity reactions to heparin and synthetic oligosaccharides. Thromb Haemost. 2005 Dec;94(6):1265-9. doi: 10.1160/TH05-05-0318. PMID 16411404
- [Background] Warkentin TE, Roberts RS, Hirsh J, Kelton JG. Heparin-induced skin lesions and other unusual sequelae of the heparin-induced thrombocytopenia syndrome: a nested cohort study. Chest. 2005 May;127(5):1857-61. doi: 10.1378/chest.127.5.1857. PMID 15888871
- [Background] Maetzke J, Hinrichs R, Schneider LA, Scharffetter-Kochanek K. Unexpected delayed-type hypersensitivity skin reactions to the ultra-low-molecular-weight heparin fondaparinux. Allergy. 2005 Mar;60(3):413-5. doi: 10.1111/j.1398-9995.2005.00695.x. No abstract available. PMID 15679737
- [Background] Gaigl Z, Pfeuffer P, Raith P, Brocker EB, Trautmann A. Tolerance to intravenous heparin in patients with delayed-type hypersensitivity to heparins: a prospective study. Br J Haematol. 2005 Feb;128(3):389-92. doi: 10.1111/j.1365-2141.2004.05321.x. PMID 15667543
- [Background] Hirsch K, Ludwig RJ, Lindhoff-Last E, Kaufmann R, Boehncke WH. Intolerance of fondaparinux in a patient allergic to heparins. Contact Dermatitis. 2004 Jun;50(6):383-4. doi: 10.1111/j.0105-1873.2004.0350j.x. No abstract available. PMID 15274739
- [Background] Koch P. Delayed-type hypersensitivity skin reactions due to heparins and heparinoids. Tolerance of recombinant hirudins and of the new synthetic anticoagulant fondaparinux. Contact Dermatitis. 2003 Dec;49(6):276-80. doi: 10.1111/j.0105-1873.2003.0255.x. PMID 15025697
- [Background] Ludwig RJ, Beier C, Lindhoff-Last E, Kaufmann R, Boehncke WH. Tolerance of fondaparinux in a patient allergic to heparins and other glycosaminoglycans. Contact Dermatitis. 2003 Sep;49(3):158-9. doi: 10.1111/j.0105-1873.2003.0185a.x. No abstract available. PMID 14678213
- [Background] Warkentin TE, Sheppard JA, Sigouin CS, Kohlmann T, Eichler P, Greinacher A. Gender imbalance and risk factor interactions in heparin-induced thrombocytopenia. Blood. 2006 Nov 1;108(9):2937-41. doi: 10.1182/blood-2005-11-012450. Epub 2006 Jul 20. PMID 16857993
- [Derived] Schindewolf M, Scheuermann J, Kroll H, Marzi I, Kaufmann R, Boehncke WH, Ludwig RJ, Lindhoff-Last E. Application, tolerance and safety of fondaparinux therapy in a German hospital: a prospective single-centre experience. Thromb Res. 2012 Jan;129(1):17-21. doi: 10.1016/j.thromres.2011.06.008. Epub 2011 Jul 7. PMID 21741076
- [Derived] Schindewolf M, Scheuermann J, Kroll H, Garbaraviciene J, Hecking C, Marzi I, Wolter M, Kaufmann R, Boehncke WH, Lindhoff-Last E, Ludwig RJ. Low allergenic potential with fondaparinux: results of a prospective investigation. Mayo Clin Proc. 2010 Oct;85(10):913-9. doi: 10.4065/mcp.2010.0346. Epub 2010 Sep 15. PMID 20843983
- [Derived] Schindewolf M, Schwaner S, Wolter M, Kroll H, Recke A, Kaufmann R, Boehncke WH, Lindhoff-Last E, Ludwig RJ. Incidence and causes of heparin-induced skin lesions. CMAJ. 2009 Oct 13;181(8):477-81. doi: 10.1503/cmaj.081729. Epub 2009 Sep 28. PMID 19786468
- See also: Homepage of the Department of Internal Medicine (Angiology) with contact persons in the angiology department listed (site in German) — http://www.gefaesszentrum-frankfurt.de